CLINICAL TRIAL: NCT04377841
Title: Clinical Correlation Between Facial Demodicosis and Ocular Demodicosis
Brief Title: Facial Demodicosis and Ocular Demodicosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201912024RIND
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Demodex Infestation; Rosacea; Blepharitis; Meibomian Gland Dysfunction; Pityriasis Folliculorum
Keywords: Demodex; Facial Demodicosis; Ocular Demodicosis; Direct Microscopic Examination; Rosacea; Blepharitis; Meibomian Gland Dysfunction; Pityriasis Folliculorum
MeSH Terms: conditions — Rosacea; Blepharitis; Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Facial Demodicosis: 1. Clinical presentation of facial skin matches any of the followings:
     1. Pityriasis folliculorum.
     2. Papulopustular lesion.
     3. Rosacea.
  2. Demodex infestation detected by direct microscopic examination ≥ 5 mites/cm2.
- Ocular Demodicosis: 1. Clinical presentation of ocular region matches any of the followings:
     1. Chronic blepharitis.
     2. Eyelash abnormalities: trichiasis, distichiasis, madarosis.
     3. Meibomian gland dysfunction.
     4. Recurrent chalazion.
     5. Ocular rosacea.
  2. Demodex infestation detected by cilia epilation test ≥ 1 mite/eyelid.

SUMMARY:
To understand the association between facial demodicosis and ocular demodicosis, we plan to enroll patients with facial demodicosis, ocular demodicosis, or both, in order to analyze their clinical presentations, the density of Demodex infestation over facial skin and eyelashes, and possible risk factors of the two diagnoses.

DETAILED DESCRIPTION:
Although facial demodicosis and ocular demodicosis are described in a variety of clinical presentations, the association between the two diagnoses is not clearly identified.

Clinically, we plan to enroll 120 patients with facial demodicosis, ocular demodicosis. We will obtain their basic information, medical history, medication, and lifestyle. We will evaluate their clinical features. We will also perform quantitative tests including direct microscopic examination and cilia epilation test:

1. Direct microscopic examination: On glabella and bilateral cheeks, follicular contents in the 1-cm × 1-cm area will be squeezed out. The contents are transferred onto a glass slide, covered with mineral oil and a cover slide, and examined under the microscope.
2. Epilation: Four (4) non-adjacent cilia will be pulled from each upper eyelid and examined under the microscope. The total Demodex counts are recorded.

We will analyze the clinical presentations, the density of Demodex infestation, and possible risk factors of the two diagnoses.

ELIGIBILITY:
Inclusion Criteria:

Patient with a diagnosis of facial demodicosis or ocular demodicosis.

A. Facial demodicosis defined as both 1 and 2:

1. Clinical presentation of facial skin matches any of the followings:

   1. Pityriasis folliculorum.
   2. Papulopustular lesion.
   3. Rosacea.
2. Demodex infestation detected by direct microscopic examination ≥ 5 mites/cm2.

   B. Ocular demodicosis defined as both 3 and 4:
3. Clinical presentation of ocular region matches any of the followings:

   1. Chronic blepharitis.
   2. Eyelash abnormalities: trichiasis, distichiasis, madarosis.
   3. Meibomian gland dysfunction.
   4. Recurrent chalazion.
   5. Ocular rosacea.
4. Demodex infestation detected by cilia epilation test ≥ 1 mite/eyelid.

Exclusion Criteria:

1. Usage of oral Ivermectin, topical Ivermectin or topical tea tree oil in the past 1 month.
2. Patient who cannot tolerate direct microscopic examination or cilia epilation test.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 years or older and with a diagnosis of either facial demodicosis or ocular demodicosis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-12-14 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
Quantitative tests of facial and ocular demodicosis | On initial evaluation
  Association between the results of direct microscopic examination and cilia epilation test

SECONDARY OUTCOMES:
Clinical features and quantitative tests of facial demodicosis | On initial evaluation
  Association between the clinical features and the result of direct microscopic examination
Clinical features and quantitative tests of ocular demodicosis | On initial evaluation
  Association between the clinical features and the result of cilia epilation

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Plewig G. Human demodicosis: revisit and a proposed classification. Br J Dermatol. 2014 Jun;170(6):1219-25. doi: 10.1111/bjd.12850. PMID 24471456
- [Background] Askin U, Seckin D. Comparison of the two techniques for measurement of the density of Demodex folliculorum: standardized skin surface biopsy and direct microscopic examination. Br J Dermatol. 2010 May;162(5):1124-6. doi: 10.1111/j.1365-2133.2010.09645.x. Epub 2010 Feb 25. PMID 20199545
- [Background] Gao YY, Di Pascuale MA, Li W, Liu DT, Baradaran-Rafii A, Elizondo A, Kawakita T, Raju VK, Tseng SC. High prevalence of Demodex in eyelashes with cylindrical dandruff. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3089-94. doi: 10.1167/iovs.05-0275. PMID 16123406